CLINICAL TRIAL: NCT05396651
Title: Effect of Low Fodmap Diet on Control of Pediatric Irritable Bowel Syndrome
Brief Title: Effect of Low Fermentable Oligosaccharides, Disaccharides ,Monosaccharides and Polyols (FODMAP) Diet on Control of Pediatric Irritable Bowel Syndrome and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Abdelrahman El Ezaby (Other)
Responsible Party: Sponsor-Investigator, Sarah Abdelrahman El Ezaby, Family Medicine assistant lecturer at Faculty of Medicine, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU319/2019
Record Dates: First submitted 2022-03-06; First posted 2022-05-31 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOW FODMAP Diet group (Experimental): 42 Children aged 5-15 years old fulfilling ROME IV criteria of IBS diagnosis, and didn't have any of the following :o Abdominal pain or diarrhea that wakes the child from sleep
  * Delay in onset or progression of puberty.
  * Faltering growth.
  * Family history of inflammatory bowel disease, celiac disease.
  * History of significant weight loss .
  * Bleeding per rectum.
  * Persistence of severe vomiting or diarrhea
  * . Persistent joint pain.
  * Recurrent unexplained fever.
  * Unexplained pallor they followed the low fodmapdiet for 6 weeks
  Interventions: Other: low fodmap diet
- NICE guidelines group (Placebo Comparator): 42 Children aged 5-15 years old fulfilling ROME IV criteria of IBS diagnosis and didn't have one of the following : o Abdominal pain or diarrhea that wakes the child from sleep
  * Delay in onset or progression of puberty.
  * Faltering growth.
  * Family history of inflammatory bowel disease, celiac disease.
  * History of significant weight loss .
  * Bleeding per rectum.
  * Persistence of severe vomiting or diarrhea
  * . Persistent joint pain.
  * Recurrent unexplained fever.
  * Unexplained pallor
  they followed NICE guidelines for irritable bowel syndrome for 6 weeks
  Interventions: Other: NICE guidelines for IBS

INTERVENTIONS:
Other: low fodmap diet — elimination of high fodmap diet - High FODMAP diet: ice cream, soft cheese , yoghurt, cabbage , cauliflower, green bean, garlic, okra, onions, snow peas, broccoli, avocado , apple, mango , dates, watermelon, legumes , pulses, wheat , pasta , artificial sweeteners
  Arms: LOW FODMAP Diet group
Other: NICE guidelines for IBS — follow NICE guidelines for IBS :have regular meals and take time to eat. avoid missing meals or leaving long gaps between eating. drink at least 8 cups of fluid per day, especially water or other non-caffeinated drinks, for example herbal teas.
  restrict tea and coffee to 3 cups per day. reduce intake of alcohol and fizzy drinks.
  Arms: NICE guidelines group

SUMMARY:
To evaluate the impact of low FODMAP diet on Health related Quality of life in children with Irritable bowel syndrome according to ROME IV criteria in a group of patients in pediatric Hospital at Ain Shams University

DETAILED DESCRIPTION:
Single blinded randomized two-arm intervention study in which 42 patients with irritable bowel syndrome were enrolled to study the effect of LOW FODMAP diet ( intervention group) on their gastrointestinal symptoms and their quality of life another group of 42 patients of IBS were enrolled as a control group who were received general diet instructions and they followed the NICE guide lines for IBS management

ELIGIBILITY:
Inclusion Criteria:

* children aged 5-15 years old fulfilling ROME IV criteria of IBS diagnosis

Exclusion Criteria:

Patients presenting with :

* Abdominal pain or diarrhea that wakes the child from sleep
* Delay in onset or progression of puberty.
* Faltering growth.
* Family history of inflammatory bowel disease, celiac disease.
* History of significant weight loss .
* Bleeding per rectum.
* Persistence of severe vomiting or diarrhea
* . Persistent joint pain.
* Recurrent unexplained fever.
* Unexplained pallor

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
improvement of irritable bowel syndrome symproms | 6 weeks
  Change in Pediactric Quality of life inventory (PedsQL) gastrointestinal symptoms module score

SECONDARY OUTCOMES:
improve patients quality of life | 6 weeks
  Change in Pediatric quality of life inventory (PEDSQL) Generic core l score

CONTACTS AND LOCATIONS:
Overall Officials: Diaa a Marzouk, professor, Study Director — faculty of medicine ain shams university
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No